CLINICAL TRIAL: NCT05230459
Title: A Two-part Multicenter Study: a Randomized, Double-blind, Placebo-controlled Dose-escalation Safety Phase (Part 1) Followed by Double-blind, Placebo-controlled, Adaptive Phase (Part 2) Study to Evaluate the Safety and Efficacy of AB-1003 in Adult Subjects With LGMD2I/R9 Mutations in the Gene Encoding Fukutin Related Protein (FKRP)
Brief Title: A Study to Evaluate the Safety of AB-1003 (Previously LION-101) in Subjects With Genetic Confirmation of LGMD2I/R9 (Part1)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AskBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LION-CS101
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Limb Girdle Muscular Dystrophy; Limb-Girdle Muscular Dystrophy Type 2; LGMD2I; Muscular Dystrophy; LGMD2; LGMD; FKRP; FKRP Mutation; Fukutin Related Protein
Keywords: gene therapy; LGMD2I; LGMD2I/R9; gene augmentation therapy; FKRP; fukutin related protein; FKRP mutation
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle; Limb-girdle muscular dystrophy type 2A; Muscular Dystrophy, Limb-Girdle, Type 2I; Muscular Dystrophies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AB-1003 Cohort 1 (Experimental)
  Interventions: Genetic: AB-1003 dose level 1
- AB-1003 Cohort 2 (Experimental)
  Interventions: Genetic: AB-1003 dose level 2
- Placebo (Cohorts 1 and 2) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Genetic: AB-1003 dose level 1 — Single intravenous infusion of AB-1003 gene therapy at dose level 1
  Arms: AB-1003 Cohort 1
Genetic: AB-1003 dose level 2 — Single intravenous infusion of AB-1003 gene therapy at dose level 2
  Arms: AB-1003 Cohort 2
Other: Placebo — Single intravenous infusion of Placebo
  Arms: Placebo (Cohorts 1 and 2)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a single intravenous infusion of AB-1003 in adults diagnosed with limb girdle muscular dystrophy type 2I/R9 (LGMD2I/R9). Participants will be treated in sequential, dose-level cohorts. (Part 1)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 and 65 years with clinical diagnosis of LGMD2I/R9 and confirmation of FKRP gene mutation.
2. Ability to ascend 4 stairs between 2.5 and 10 seconds.
3. Ability to walk/run 10 meters in <30 seconds.
4. Able to understand and comply with all study procedures.
5. Sexually active females of childbearing potential and female and male partners of male subjects receiving study intervention must use a barrier method of contraception for the first 6 months after dosing.

Exclusion Criteria:

1. Significant cardiomyopathy as defined by echocardiogram (left ventricular ejection fraction <40%), evidence of conduction defect (increased PR and RR intervals, left bundle branch block and QTcF >480m/sec), NYHA Class 3 or 4 heart failure, or MRI gadolinium enhancement evidence of clinically important myocardial fibrosis.
2. Contraindication to MRI or hypersensitivity to contrast dyes, shellfish or iodine.
3. Implanted spinal rods, cardiac pacemaker or other implantation that would distort cardiac MRI images.
4. History of active, ongoing chronic liver disease (e.g. hepatitis, HIV-related liver disease, hemochromatosis, steatosis, etc.) or abnormal liver function tests (abnormal GGT and/or abnormal total/direct bilirubin >upper limit of normal [ULN] and/or elevated AST and ALT >2 ULN).
5. Abnormal renal function (GFR <60 ml/min, using the Modification of Diet in Renal Disease equation).
6. Any life-threatening disease, including malignant neoplasms and medical history or malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
7. In the opinion of the investigator, a pre-existing medical condition that predisposes the subject to risks that outweighs the potential benefits.
8. Requirement for daytime ventilatory support.
9. Change in glucocorticosteroid treatment within 3 months prior to screening visit.
10. Exposure to another investigational drug within 3 months prior to study treatment or any previous treatment with gene therapy.
11. Ongoing participation in any other therapeutic clinical trial.
12. Neutralizing antibody titer to AAV9 >1:5.
13. Female subjects who are pregnant, plan to become pregnant in the next 12 months, or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 0-52 weeks
  Treatment Emergent Adverse Events, Serious Adverse Events, Dose Limiting Toxicity

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California - Irvine, Irvine, California
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - VCU, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to webpage for study and pre-qualification information — https://mytomorro.ws/lion-101-gov